CLINICAL TRIAL: NCT01741428
Title: "Hjerteloeftet". Early Interventions to Promote Physical Activity, Dietary Lifestyle Changes and Optimal Medication for Cardiovascular Risk Factor Reduction in Over 3 Years Follow-up.
Brief Title: "Hjerteloeftet" ("HeartLift"). Interaction For Preventing Cardiovascular Disease
Acronym: HeartLift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011/561a(REK-LHL)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Disease
Keywords: CVD Risk score; Physical activity; Overweight; Cholesterol; LDL-Cholesterol; HDL-Cholesterol; Triglycerides; HbA1C; Quality of life
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Overweight | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intervention (INT1) (Active Comparator): The participants will join a 5-days course at the Feiring Heart Clinic.
  Interventions: Behavioral: Intervention (INT1)
- Control (KTR1) (No Intervention): The participants in the Control Group will receive care as usual at their local Doctors Office
- Subgroup Intervention (INT2) (Active Comparator): Subgroup of 200 participants from the (INT1)where multiple, known CVD risk factors are studied: Physical Activity, Physical Condition (O2-consumption), Quality of life, Biochemical markers (fasting Glucose, Insulin, Apo Lipoprotein A (ApoA), Apo Lipoprotein B (ApoB), micro-C reactive protein (CRP), Total-, LDL- and HDL-cholesterol, Triglycerides and HbA1C.
  Interventions: Behavioral: Intervention (INT1)
- Subgroup control (KTR2) (No Intervention): Subgroup of 200 participants from the (KTR1)where multiple, known CVD risk factors are studied: Physical Activity, Physical Condition (O2-consumption), Quality of life, Biochemical markers (fasting Glucose, Insulin, Apo Lipoprotein A (ApoA), Apo Lipoprotein B (ApoB), micro-C reactive protein (CRP), Total-, LDL- and HDL-cholesterol, Triglycerides and HbA1C.

INTERVENTIONS:
Behavioral: Intervention (INT1) — The course Program at the Feiring Heart Clinic will:
  Clinical examination and ergospirometric testing, optimizing both treatment and prophylactic medication. Promoting physical Activity, changes in lifestyle, dietary changes/weight reduction, smoking cessation. In the follow-up period the participants will be contacted and report regularly through a web-based secure program (MedAxess)(such as: Activity-, dietary- and smoking habits). Each participant will have their own Mentor, helping keeping up the motivation. They will also meet regularly at the local doctors Office which reports relevant parameters to the Project (such as weight, BP, Lipoproteins, blood glucose/HbA1C)
  Arms: Intervention (INT1); Subgroup Intervention (INT2)

SUMMARY:
Early interventions to promote physical activity, dietary lifestyle changes and optimal medication for cardiovascular risk factor reduction - 3 years follow-up. A randomized Clinical Trial.

DETAILED DESCRIPTION:
Background

It has been established that the major risk factors of coronary artery disease are modifiable risk factors. The international Case control study across 52 countries has identified that 90% of the risk of acute myocardial infarction in males and 94% in females were modifiable risk factors as smoking habits, presence of hypertension, diabetes mellitus, abdominal obesity, psychological and social stress and hyperlipidemia (1).

It is well established that interventions to promote physical activity and dietary changes could have beneficial effect in the reduction of incidence of coronary heart disease (CHD) (2).

Aim of the Study

The research hypothesis is that for persons on medium to high risk of CHD an early intervention using lifestyle and drugs over a period of three years can reduce the patients risk to develop CHD as estimated by risk score and some established risk factors of CHD as secondary surrogate end points.

Major End Point

For the major end point change in NORRISK Score (3) a systematic review of the literature to estimate sample size for a power estimate was done in association with a pilot study to estimate the variability of the score. The outcome variable is difference in risk score between baseline and three years follow-up. Considering the analysis of the pilot study, the investigators estimated the variability of the score difference (delta) of NORRISK to be standard deviation = 6.18%. As the median age of this sample was 51 years it is considered a change in the probability of ten years cardiovascular death of 1.5% to be clinically interesting. For a power of 90% and a type-I error of 5% the study will need two times 358 patients. Accepting a 10% dropout in the actual population, the corrected sample size will be two times 394. A total of 800 patients, two times 400, could be enough to pinpoint substantial risk change between baseline and three years follow-up for the NORRISK score.

Secondary end points

The investigators have done an extensive research of the literature as far the effect of lifestyle intervention on different surrogate end points as change in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP), weight in kg, change in waist circumference in cm and change in TG, HDL-, LDL- Cholesterol, and HBA1C. (4, 5, 6).

From the literature the estimated change between baseline and one year of intervention are:

1. Change in weight for the intervention is - 4.2kg (SD=5.1) and in percent - 4.75 % (SD=5.4). For the control group it is - 0.8 kg (SD=3.7) and - 0.9% (SD=4.2).
2. Change in waist circumference in cm for the intervention is - 4.4 cm (SD=5.2) for the control - 1.3 cm (SD=4.8).
3. Change in serum lipid in mg/dl:

Cholesterol mg/dl for the intervention - 5mg/dl (SD=2.8) for the control - 1.3 mg/dl (SD=2.8) HDL in mg/dl for the intervention 2 mg/dl (SD=7) for the control 1 mg/dl (SD=6) TG in mg/dl for the intervention -18 mg/dl (SD=51) and intervention -1 mg/dl (SD=60) d) Change in BMI in percent after one year for the intervention group -6.7% and the control -1.4% according to (6))

Considering those figure from the literature for a power of 80% and a type - I error of 5% the investigators will need the following minimum sample size:

* Change in weight in kg 2*27 = 54 patients, in percent 2*48 = 96 patients
* Change in SBP and DBP in mmHg:

SBP mmg 2*207 = 414 patients DBP mmg 2*318 = 636 patients

* Change in BMI in percent 2*214 = 428 patients
* Changes in Triglycerides (TG) 2*169 = 338 patients

In this clinical trial there will surely be enough power with a sample size of' 2*220 = 440 patients for the major surrogate outcomes except for changes in Cholesterol and HDL. As the intervention time is longer than three years instead of one year, those power estimates could under estimate the "de facto" power at the end of the three years observation time.

Study population

Selection criteria

All persons who are selected from the general practitioner physician (GP) offices in all Norway. This study use the NORRISK Score (3), a new guideline for prevention of CardioVascular Disease (CVD) that includes calculation of total risk. This new risk model based on updated Norwegian data, as the European SCORE function, overestimates the risk of fatal CVD in Norway. NORRISK for 10-year CVD mortality is presented. It includes gender, age, smoking and levels of systolic blood pressure and serum total Cholesterol.

Ten - year risk estimates calculated from NORRISK fall between SCORE high- and low risk estimates and increase strongly with age. Very few persons below 50 years of age have a 10 - year risk above 5% (European limit for high risk). More than half of men aged 60 years have estimated risks above this limit, while only 7% of 60-year-old women exceed the limit. Even if the risk limit is reduced to 1% for younger age groups, very few women below 50 years of age have risks above the limit.

NORRISK is more adapted to the current situation in Norway than the SCORE model and may be a useful and relevant tool in Norwegian clinical practice.

Randomization procedure

Patients will be randomized to intervention or usual care. Randomization will be in permuted block randomization with utilization of concealed opaque envelopes.

Patient information

At randomization the patient receives verbal and written information about the study. This information will be repeated verbally. The patients sign a formula "Consent to participate".

Ethics Committee

The committee may look into the database during the study to assess data quality and to evaluate the quality of end points. If necessary the inclusion period or follow up time could be prolonged.

Recording of data

All case report forms (CRF) will be kept for the analysis in Feiring Heart Clinic before their introduction to the database electronically.

Evaluation of data

All CRF's are checked centrally for validity and completeness.

Disclosure of data and publication

All information obtained as a result of the study will be regarded confidential until appropriate analysis and review is performed. The results will be published and presented internationally. As far authorship and contribution, the investigators will follow the recommendations from the International Committee of Medical Journal Editor (ICMJE)(www.ICMJE.org). After publication of the initial report, participating investigators may prepare and publish sub analysis. All sub studies must be approved by the steering committee. All participant investigators will be acknowledged by name in the main publication.The recommendations of the STROBE group will be followed all the way (7).

Insurance

All patients participating in the study are insured in accordance with the official Norwegian insurance regulations.

End point and adverse events review committee

* Per Mølstad, MD, Philosophiae doctor (PhD), Department of cardiology, Feiring Heart Clinic
* Dag Elle Rivrud, MD, Feiring Heart Clinic

Start and end of study

Start of study on November 25. 2012 and continue throughout 2021.

Administrative matters

A. Principal/Chief investigator

- Hilde Bergum, MD, LHL-Hospital Gardermoen

B. Steering Committee

* Siri Skumlien, Managing Director, LHL-Hospital Gardermoen
* Nils Erling Myhr, Department Head of Rehabilitation, LHL-Hospital Gardermoen
* Jostein Grimsmo, MD, PhD, Chief Med Doctor of the Rehab.Dep., LHL-Hospital Gardermoen

C. Reference Committee

* Henning Ringlund, Participant representative
* Tor Ole Klemsdal, MD, PhD, Leader of section of preventive cardiology. Center for preventive medicine, Oslo University Hospital, Ullevål.
* Sigmund Alfred Andersen, Ph.D, Professor, Norwegian School of Sport Sciences
* Per Mølstad, MD, PhD, Department of cardiology, LHL-Hospital Gardermoen
* Sigurd Kjørstad Fjeldbo, Viberg Legesenter, Smed Hagens veg 11, 2080 Eidsvoll
* Anne Marie Aas, PhD, Researcher, Clinical nutritionist Oslo University Hospital, Aker

D. Advisor(s)/Consultant(s) for research and statistical methodology

- Irene Sandven, MPH, Ph.D, Researcher, Oslo Center of biostatistics and epidemiology, Oslo University Hospital, Ullevål.

ELIGIBILITY:
Inclusion Criteria: All male and female between the age of 35 to 67 with middle or high 10 years risk estimate are included.

* >= 0.5% for persons under the age of 50 years
* >= 2.5% for persons between 50-59 years
* >= 5% for persons > 60 years

Exclusion Criteria:

* Previous cardiovascular disease (CHD ; peripherical atherosclerosis, deep venous thrombosis /pulmonary embolism, congenital heart disease, presence of valvular heart disease).
* Lung disease restricting usual physical activity .
* Serious psychological problems (that hinders the participation in the study)
* All kind of disease restricting performing adequate physical activity .
* Presence of cancer shortening drastically survival.

Ages: 35 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2012-11; Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Change in risk score (NORRISK) | 3 Years after end of inclusion
  Major End Point
  Change in risk score (Norrisk, Procam and Framingham) between baseline and after three years of intervention.

SECONDARY OUTCOMES:
Weight and Body Mass Index (BMI) | 3 Years after end of inclusion
  Change of weight in kg and BMI between baseline and three years of follow-up.
Waist circumference | 3 Years after end of inclusion
  Change of waist circumference in cm. between baseline and three years of follow-up.
Serum Lipids | 3 Years after end of inclusion
  Change of serum Lipids in mmol/l (LDL-, HDL-, Total-Cholesterol and Triglycerides) between baseline and three years of follow-up.
Blood Pressure | 3 Years after end of inclusion
  Change of Blood Pressure in mmHG between baseline and three years of follow-up.
HbA1C | 3 Years after end of inclusion
  Change of HbA1C in % between baseline and three years of follow-up.

OTHER OUTCOMES:
Interaction outcome | 3 Years after end of inclusion
  The Interaction between primary (local) and secondary (hospital) Health Service/-care) will be evaluated through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Bergum, MD, Principal Investigator — LHL Hospital Gardermoen
Locations (1):
- LHL-Hospital Gardermoen, Jessheim, Norway

REFERENCES:
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Artinian NT, Fletcher GF, Mozaffarian D, Kris-Etherton P, Van Horn L, Lichtenstein AH, Kumanyika S, Kraus WE, Fleg JL, Redeker NS, Meininger JC, Banks J, Stuart-Shor EM, Fletcher BJ, Miller TD, Hughes S, Braun LT, Kopin LA, Berra K, Hayman LL, Ewing LJ, Ades PA, Durstine JL, Houston-Miller N, Burke LE; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing. Interventions to promote physical activity and dietary lifestyle changes for cardiovascular risk factor reduction in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 27;122(4):406-41. doi: 10.1161/CIR.0b013e3181e8edf1. Epub 2010 Jul 12. No abstract available. PMID 20625115
- [Background] Selmer R, Lindman AS, Tverdal A, Pedersen JI, Njolstad I, Veierod MB. [Model for estimation of cardiovascular risk in Norway]. Tidsskr Nor Laegeforen. 2008 Jan 31;128(3):286-90. Norwegian. PMID 18264151
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Mattila R, Malmivaara A, Kastarinen M, Kivela SL, Nissinen A. Effectiveness of multidisciplinary lifestyle intervention for hypertension: a randomised controlled trial. J Hum Hypertens. 2003 Mar;17(3):199-205. doi: 10.1038/sj.jhh.1001531. PMID 12624611
- [Background] Ackermann RT, Finch EA, Brizendine E, Zhou H, Marrero DG. Translating the Diabetes Prevention Program into the community. The DEPLOY Pilot Study. Am J Prev Med. 2008 Oct;35(4):357-63. doi: 10.1016/j.amepre.2008.06.035. PMID 18779029
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- [Derived] Bergum H, Grimsmo J, Anderssen SA, Klemsdal TO. Effects on physical activity, physical fitness and well-being in a 36-months randomized controlled study, comparing a multimodal hospital-based intervention programme for primary cardiovascular prevention with usual care. BMC Cardiovasc Disord. 2024 Apr 25;24(1):225. doi: 10.1186/s12872-024-03892-1. PMID 38664620
- [Derived] Bergum H, Sandven I, Abdelnoor M, Anderssen SA, Grimsmo J, Rivrud DE, Myhr NE, Vold MB, Stenbakken C, Lidfors B, Dufseth L, Klemsdal TO. Randomized trial of cardiovascular prevention in Norway combining an in-hospital lifestyle course with primary care follow-up: the Hjerteloftet study. Eur J Prev Cardiol. 2022 Dec 7;29(17):2252-2263. doi: 10.1093/eurjpc/zwac211. PMID 36124709